CLINICAL TRIAL: NCT05642962
Title: A Randomized Double Blind Study of Pancreatic Enzyme Replacement Therapy for Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Pancrelipase in People With Pancreatic Ductal Adenocarcinoma (PDAC)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-419
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Cancer; Metastatic Pancreatic Adenocarcinoma; Metastatic Pancreatic Carcinoma; Pancreatic Carcinoma; Pancreatic Carcinoma Metastatic; Pancreatic Carcinoma Non-resectable; Pancreatic Cancer; Pancreatic Cancer Non-resectable; Pancreatic Cancer Stage IV; Pancreatic Cancer Metastatic; PDAC; PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: Metastatic Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Cancer; Pancrelipase; Memorial Sloan Kettering Cancer Center; 21-419
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants with stage 4 Pancreatic Ductal Adenocarcinoma / PDAC will receive 384 units lipase/kg of body weight per meal or snack
  Interventions: Drug: Pertzye
- Arm 2 (Experimental): Participants with stage 4 Pancreatic Ductal Adenocarcinoma / PDAC will receive 1350 units lipase/kg of body weight per meal or snack
  Interventions: Drug: Pertzye

INTERVENTIONS:
Drug: Pertzye — Treatment with standard dose or higher dose Pancrelipase will continue for 20 weeks from enrollment. Participants will consume assigned blinded weight based Pancrelipase dose concurrent with first bite of every meal and snack for the duration of enrollment.
  Other Names: Pancrelipase

SUMMARY:
The main purpose of this study is to see how pancrelipase affects the body mass index (BMI) in people with metastatic PDAC. BMI is a measure based on a person's height and weight. Other study goals are to explore two different dosing schedules of pancrelipase and to evaluate pancrelipase in people who do not have symptoms of EPI.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic or cytologic diagnosis of pancreatic adenocarcinoma, or adenosquamous cancer, or any non-neuroendocrine primary pancreas variant, including acinar cancer.
* De novo or recurrent diagnosis of previously untreated stage IV PDAC with intent to receive FOLFIRINOX/mFOLFIRINOX.
* ECOG 0-2.
* No use of pancreatic enzyme replacement therapy within prior 2 weeks.
* Patients with biliary obstruction are eligible provided biliary stenting has or will occur before treatment with FOLFIRINOX.
* Ability to understand and the willingness to sign an informed consent document.
* Ability to swallow capsules.
* Age ≥18 years.
* Anticipated life expectancy of at least 6 months.

Exclusion Criteria:

* Chronic illness associated with malabsorption (celiac disease, cystic fibrosis, chronic pancreatitis, Crohn's disease).
* Fibrosing colonopathy.
* Prior history of surgical resection of the pancreas or gastric bypass.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Pancrelipase.
* Patients cannot receive radiation, IRE, or other localized therapy directed to the pancreas while on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index/BMI from baseline to 4 months | 4 months
  The primary objective is a change in body mass index (BMI) 4 months from baseline while on pancreatic enzyme replacement therapy (PERT).

CONTACTS AND LOCATIONS:
Overall Officials: Eileen O'Reilly, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org